CLINICAL TRIAL: NCT00725452
Title: Real Life Treatment Regimen of Remicade (Infliximab) in Austria, Monitored Over 5 Years in Plaque Psoriasis Therapy
Brief Title: Five-Year Observation of Remicade Treatment for Plaque Psoriasis in Austria (Study P04900)
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Centocor, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: P04900
Record Dates: First submitted 2008-07-25; First posted 2008-07-30 (Estimated); Results first posted 2011-09-02 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Infliximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Infliximab: Subjects with plaque psoriasis will receive Infliximab initial induction therapy consisting of 3 Infliximab infusions at weeks 0, 2, and 6 given in specialized centers. A maximum of 6 maintenance infusions will be given in doses and intervals due to the discretion of the physicians.
  Interventions: Biological: Infliximab

INTERVENTIONS:
Biological: Infliximab — Infliximab initial induction therapy consisting of 3 Infliximab infusions at weeks 0, 2, and 6 given in specialized centers. A maximum of 6 maintenance infusions will be given in doses and intervals due to the discretion of the physicians.
  Other Names: Remicade; SCH 215596

SUMMARY:
Prospective, open-label-, 1-arm, multicenter observational study to determine the dose and interval of Infliximab infusions for subjects with plaque psoriasis.

DETAILED DESCRIPTION:
This study population was chosen from a non-probability sample.

ELIGIBILITY:
Inclusion Criteria:

* According to the European Summary of Product Characteristics (SPC): Adult subjects with moderate-to-severe plaque psoriasis who failed to respond to, or who have a contraindication to, or are intolerant to other systematic therapy including cyclosporine, methotrexate, or Psoralen-ultraviolet-A light (PUVA).

Exclusion Criteria:

* According to the European SPC:

  * Subjects with tuberculosis or other severe infections such as sepsis, abscesses, and opportunistic infections.
  * Subjects with moderate-to-severe heart failure (New York Heart Association (NYHA) class III/IV).
  * Subjects with a history of hypersensitivity to Infliximab or to other murine proteins or to any of the excipients.
  * Subjects with elevated liver enzymes (>5 upper limit of normal (ULN)).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects with moderate-to-severe plaque psoriasis will receive Infliximab induction therapy in specialized centers.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2006-10; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Infliximab: Infliximab induction therapy consisted of 3 infusions (5 mg/kg) in weeks 0, 2, and 6 given in specialized centers. Maintenance therapy consisted of a maximum of 6 infusions (5 mg/kg) given in doses and intervals at the discretion of the physician.
Period: Overall Study
Arm/Group | Infliximab
Started | 26
Completed | 15 (Completed was defined as the number of participants who received 9 consecutive Infliximab infusions.)
Not Completed | 11
Not completed — Adverse Event | 3
Not completed — Lack of Efficacy | 2
Not completed — Reason not specified | 1
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 3
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Infliximab
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.23 (10.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Therapies That Were Applied as Induction, Maintenance, or Episodic Therapies After One Infusion of Infliximab
Description: The types of therapies were assessed according to the following criteria:
  Induction therapy: first infusion given at Week 0 (Baseline). Second infusion given at Week 2 (+/- 7 days). Third infusion given at Week 6 (+/- 7 days).
  Maintenance therapy: given in approximately 8-week (56-day) intervals (time window +4 weeks to -2 weeks). One infusion given out of the time window was accepted to be classified as maintenance therapy, if the remaining infusions were given within the time window (8 weeks, +4 to -2 weeks).
  Episodic Therapy: given out of time frame (> 12 weeks).
Time Frame: Maximum 2 years
Population: Infliximab-naive participants who received Infliximab during the study.
Measure: Number; unit: Therapies
Arm/Group | Infliximab
Number analyzed (Participants) | 12
Therapies
  Induction therapy | 7
  Maintenance therapy | 2
  Episodic therapy | 1
  No treatment regimen applied | 2

2. Secondary Outcome: Mean Time Interval Between Infliximab Infusions During Maintenance Treatment Following Induction Therapy
Time Frame: Maximum 2 years
Population: Infliximab-naive participants who received induction therapy and subsequent maintenance therapy with Infliximab.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Infliximab
Number analyzed (Participants) | 4
Days
  Between Infusion 3 and 4 (n=4) | 49.25 (13.50)
  Between Infusion 4 and 5 (n=4) | 57.25 (2.50)
  Between Infusion 5 and 6 (n=3) | 59.67 (8.14)
  Between Infusion 6 and 7 (n=3) | 55.00 (3.61)
  Between Infusion 7 and 8 (n=3) | 56.00 (0)
  Between Infusion 8 and 9 (n=2) | 55.50 (2.12)

3. Secondary Outcome: Median Time Interval Between Infliximab Infusions During Maintenance Treatment Following Induction Therapy
Time Frame: Maximum 2 years
Population: Infliximab-naive participants who received induction therapy and subsequent maintenance therapy with Infliximab.
Measure: Mean (Full Range); unit: Days
Arm/Group | Infliximab
Number analyzed (Participants) | 4
Days
  Between Infusion 3 and 4 (n=4) | 56.00 [29 to 56]
  Between Infusion 4 and 5 (n=4) | 56.00 [56 to 61]
  Between Infusion 5 and 6 (n=3) | 56.00 [54 to 69]
  Between Infusion 6 and 7 (n=3) | 56.00 [51 to 58]
  Between Infusion 7 and 8 (n=3) | 56.00 [56 to 56]
  Between Infusion 8 and 9 (n=2) | 55.50 [54 to 57]

4. Secondary Outcome: Mean Dose of Infliximab
Time Frame: Maximum 2 years
Population: All participants who received at least 1 Infliximab infusion during the observational phase.
Measure: Mean (Standard Deviation); unit: milligrams/kilograms (mg/kg)
Arm/Group | Infliximab
Number analyzed (Participants) | 26
milligrams/kilograms (mg/kg)
  Infusion 1 (n=26) | 4.55 (0.85)
  Infusion 2 (n=23) | 4.66 (0.89)
  Infusion 3 (n=23) | 4.67 (0.93)
  Infusion 4 (n=21) | 4.58 (0.97)
  Infusion 5 (n=18) | 4.51 (0.89)
  Infusion 6 (n=16) | 4.41 (0.91)
  Infusion 7 (n=16) | 4.44 (0.91)
  Infusion 8 (n=16) | 4.16 (1.02)
  Infusion 9 (n=14) | 4.30 (1.06)

5. Secondary Outcome: Median Dose of Infliximab
Time Frame: Maximum 2 years
Population: All participants who received at least 1 Infliximab infusion during the observational phase.
Measure: Median (Full Range); unit: mg/kg
Arm/Group | Infliximab
Number analyzed (Participants) | 26
mg/kg
  Infusion 1 (n=26) | 4.88 [2.73 to 5.31]
  Infusion 2 (n=23) | 5.00 [2.68 to 5.48]
  Infusion 3 (n=23) | 5.00 [2.61 to 5.56]
  Infusion 4 (n=21) | 5.00 [2.61 to 5.41]
  Infusion 5 (n=18) | 4.91 [2.95 to 5.23]
  Infusion 6 (n=16) | 4.71 [2.98 to 5.30]
  Infusion 7 (n=16) | 4.94 [2.98 to 5.06]
  Infusion 8 (n=16) | 4.68 [2.86 to 5.06]
  Infusion 9 (n=14) | 4.94 [2.86 to 5.06]

6. Secondary Outcome: Mean Percent Change From Baseline in Body Surface Area (BSA) Involved With Psoriasis After Treatment With Infliximab
Description: BSA estimation was determined using the participant's handprint (palmar surface of palms plus five digits). The number of handprints that covered the affected skin area was counted. One handprint was approximately equivalent to 1 percent of the BSA; therefore, BSA was calculated in percentages. The change from Baseline in BSA was calculated by subtracting Baseline from infusion 9.
Time Frame: Baseline and Infusion 9
Population: Infliximab-naive participants who received Infliximab during the study.
Measure: Mean (Standard Deviation); unit: Percent of BSA involved with psoriasis
Arm/Group | Infliximab
Number analyzed (Participants) | 8
Percent of BSA involved with psoriasis
  Baseline | 38.63 (25.63)
  Change from Baseline after Infusion 9 | -11.17 (21.22)

ADVERSE EVENTS:
Arm/Group | Infliximab
Serious Adverse Events (participants affected / at risk) | 2/26
Other Adverse Events (participants affected / at risk) | 4/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infliximab (N=26)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1)
Hospitalisation (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infliximab (N=26)
Pharyngitis (Infections and infestations) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No